CLINICAL TRIAL: NCT00719888
Title: Transplantation of Umbilical Cord Blood for Patients With Hematological Diseases With Cyclophosphamide/Fludarabine/Total Body Irradiation or Cyclophosphamide/Fludarabine/Thiotepa/Total Body Irradiation Myeloablative Preparative Regimen
Brief Title: Umbilical Cord Blood Transplant, Cyclophosphamide, Fludarabine, and Total-Body Irradiation in Treating Patients With Hematologic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Ann Dahlberg, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010.00; NCI-2010-00190 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010 (Other: Fred Hutch/University of Washington Cancer Consortium); RG2807002 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Acute Biphenotypic Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Burkitt Lymphoma; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Follicular Lymphoma; Lymphoblastic Lymphoma; Lymphoplasmacytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Non-Hodgkin Lymphoma; Plasma Cell Myeloma; Prolymphocytic Leukemia; Refractory Anemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Myelodysplastic Syndromes; Primary Myelofibrosis; Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Prolymphocytic; Anemia, Refractory | interventions — Cyclophosphamide; Cyclosporine; Cyclosporins; fludarabine; Mycophenolic Acid; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (myeloablative UCBT) (Experimental): Patients receive myeloablative conditioning comprising fludarabine IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 and -6, and undergo high-dose TBI BID on days -4 to -1. Patients then undergo single- or double-unit UCBT on day 0.
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Interventions: Drug: Cyclophosphamide; Drug: Cyclosporine; Procedure: Double-Unit Umbilical Cord Blood Transplantation; Drug: Fludarabine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation
- Arm II (myeloablative UCBT) (Experimental): Patients receive myeloablative conditioning comprising fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 2-4 hours on days -5 and -4, and middle-intensity TBI QD on days -2 and -1. Patients then undergo single- or double-unit UCBT on day 0.
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Interventions: Drug: Cyclophosphamide; Drug: Cyclosporine; Procedure: Double-Unit Umbilical Cord Blood Transplantation; Drug: Fludarabine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation; Drug: Thiotepa

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cyclosporine — Given IV and PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Procedure: Double-Unit Umbilical Cord Blood Transplantation — Undergo double-unit UCBT
Drug: Fludarabine — Given IV
  Other Names: 118218; Fluorovidarabine
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given IV and PO
  Other Names: Cellcept; MMF
Radiation: Total-Body Irradiation — Undergo high-dose or moderate-intensity TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation; SCT_TBI; TBI
Procedure: Umbilical Cord Blood Transplantation — Undergo UCBT
  Other Names: Cord Blood Transplantation; UCB transplantation
Drug: Thiotepa — Given IV
  Other Names: 1,1',1"-phosphinothioylidynetrisaziridine; 1,1',1''-Phosphinothioyldynetrisaziridine; 52-24-4; 6396; Girostan; Triethylenethiophosphoramide; Triethylene Thiophosphoramide
  Arms: Arm II (myeloablative UCBT)

SUMMARY:
This phase II trial studies how well giving an umbilical cord blood transplant together with cyclophosphamide, fludarabine, and total-body irradiation (TBI) works in treating patients with hematologic disease. Giving chemotherapy, such as cyclophosphamide and fludarabine, and TBI before a donor umbilical cord blood transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

DETAILED DESCRIPTION:
OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients receive myeloablative conditioning comprising fludarabine intravenously (IV) over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 and -6, and undergo high-dose TBI twice daily (BID) on days -4 to -1. Patients then undergo single- or double-unit UCBT on day 0.

ARM II: Patients receive myeloablative conditioning comprising fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 2-4 hours on days -5 and -4, and middle-intensity TBI once daily (QD) on days -2 and -1. Patients then undergo single- or double-unit UCBT on day 0.

Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine orally (PO) (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) three times daily (TID) on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.

After completion of study treatment, patients are followed up at 6 months, 1 year, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* GRAFT CRITERIA:

  * UCB units will be selected according to current umbilical cord blood graft selection algorithm; one or 2 UCB units may be used to achieve the required cell dose
  * The UCB graft is matched at 4-6 human leukocyte antigen (HLA)-A, B, DRB1 antigens with the recipient; this may include 0-2 antigen mismatches at the A or B or DRB1 loci; unit selection based on cryopreserved nucleated cell dose and HLA-A,B, DRB1 using intermediate resolution A, B antigen and DRB1 allele typing
  * If 2 UCB units are required to reach the target cell dose, each unit must be a 4-6 antigen match to the recipient
* Age and Disease Criteria:

  * High-dose TBI regimen: 6 months to =< 45 years
  * Middle-intensity TBI regimen: 6 months to =< 65 years
  * Conditioning regimen selection should be based on the underlying disease, presence of minimum residual disease (MRD), age, co-morbidities, and attending physician
* Acute myeloid leukemia, including biphenotypic acute leukemia or mixed-lineage leukemia:

  * All patients must be in complete remission (CR) as defined by hematologic recovery and < 5% blasts by morphology/flow cytometry in a representative bone marrow sample with cellularity >= 15% for age; patients who do not have high-risk features (for example preceding myelodysplastic syndrome [MDS], high-risk cytogenetics, >= 2 cycles to obtain CR, erythroblastic or megakaryocytic leukemia or >= CR2) must be discussed with the principal investigator (PI) prior to enrollment and at the Patient Care Conference or equivalent group such as the pediatric leukemia board as an alternative
  * Patients in whom adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures; these patients must be discussed with the PI prior to enrollment; patients persistently aplastic for greater than one month since completing last chemotherapy are also eligible with PI approval
* Very high risk pediatric/young adult patients with acute myeloid leukemia (AML): Patients =< 25 years, however, are eligible with (M2 marrow) with =< 25% blasts in marrow after having failed one or more cycles of chemotherapy; this group of patients will be analyzed separately
* Acute lymphoblastic leukemia, including biphenotypic acute leukemia or mixed-lineage leukemia:

  * All patients must be in CR as defined by < 5% blasts by morphology; flow cytometry in a representative bone marrow sample with cellularity >= 15% for age; patients who do not have high-risk disease (high risk CR1, greater than one cycle to obtain CR or >= CR2) must be discussed with the PI prior to enrollment and at the Patient Care Conference or equivalent group such as the pediatric leukemia board as an alternative
  * Patients in whom adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures; these patients must be discussed with the principal investigator Ann Dahlberg prior to enrollment; patients persistently aplastic for greater than one month since completing last chemotherapy are also eligible with PI approval
* Chronic myelogenous leukemia excluding refractory blast crisis; to be eligible in first chronic phase (CP1) patient must have failed or be intolerant to imatinib mesylate
* Advanced myelofibrosis
* Myelodysplasia (MDS) International Prognostic Scoring System (IPSS) intermediate (Int)-2 or high risk (i.e., refractory anemia with excess blasts [RAEB], RAEB in transformation [RAEBt]) or refractory anemia with severe pancytopenia or high risk cytogenetics; blasts must be < 10% by a representative bone marrow aspirate morphology
* Lymphoblastic lymphoma, Burkitt's lymphoma, and other high-grade non-Hodgkin lymphoma (NHL) after initial therapy if stage III/IV in first partial response (PR1) or after progression if stage I/II < 1 year; stage III/IV patients are eligible after progression in CR/PR
* Chronic lymphocytic leukemia /small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, lymphoplasmacytic lymphoma or follicular lymphoma that have progressed after at least two different prior therapies; patients with bulky disease (nodal mass greater than 5 cm) should be considered for debulking chemotherapy before transplant; these patients must be presented at primary care center (PCC) prior to enrollment, given potential competing eligibility on autotransplant protocols
* Mantle-cell lymphoma, prolymphocytic leukemia: Eligible after initial therapy in >= CR1 or >= PR1
* Large cell NHL > CR2/> second partial response (PR2):

  * Patients in CR2/PR2 with initial short remission (< 6 months) are eligible
  * These patients must be presented at PCC prior to enrollment, given potential competing eligibility on autotransplant protocols
* Multiple myeloma beyond PR2: Patients with chromosome 13 abnormalities, first response lasting less than 6 months, or beta-2 microglobulin > 3 mg/L, may be considered for this protocol after initial therapy
* Performance status score: Karnofsky (for adults) >= 70% or Eastern Cooperative Oncology Group (ECOG) 0-1 or Lansky (for children) >= 50%
* Creatinine < 2.0 mg/dL (for adults) or creatinine clearance > 60 ml/min (for children)
* Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, histology, and the degree of portal hypertension; patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease will be excluded
* Diffusion capacity for carbon monoxide corrected (DLCOcorr) > 50% normal or a pediatric patient who is unable to perform pulmonary function tests (PFTs) but has adequate pulmonary function
* Left ventricular ejection fraction > 45% or shortening fraction > 26%

Exclusion Criteria:

* Uncontrolled viral or bacterial infection at the time of study enrollment
* Active or recent (prior 6 month) invasive fungal infection without interdisciplinary (ID) consult and approval
* History of human immunodeficiency virus (HIV) infection
* Pregnant or breastfeeding
* Chemotherapy refractory large cell and high grade NHL (i.e., progressive disease after > 2 salvage regimens)
* Patients with history of prior myeloablative transplant containing full dose TBI (greater than 8 gray [Gy]) will not be eligible for Regimen A; however, they may still enroll on Regimen B if they otherwise meet inclusion and exclusion criteria
* Any prior myeloablative transplant within the last 6 months
* Patients >= 45 years: comorbidity score of 5 or higher
* Patients who have received Y-90 ibritumomab (Zevalin) or I-131 tostumomab (Bexxar), as part of their salvage therapy are not eligible for Regimen A

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2005-11-18 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann E. Dahlberg, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide: Patients receive myeloablative conditioning comprising fludarabine IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 and -6, and undergo high-dose TBI BID on days -4 to -1. Patients then undergo single- or double-unit UCBT on day 0.
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Cyclophosphamide: Given IV
  Cyclosporine: Given IV and PO
  Double-Unit Umbilical Cord Blood Transplantation: Undergo double-unit UCBT
  Fludarabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV and PO
  Total-Body Irradiation: Undergo high-dose or moderate-intensity TBI
  Umbilical Cord Blood Transplantation: Undergo UCBT
- Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa: Patients receive myeloablative conditioning comprising fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 2-4 hours on days -5 and -4, and middle-intensity TBI QD on days -2 and -1. Patients then undergo single- or double-unit UCBT on day 0.
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Cyclophosphamide: Given IV
  Cyclosporine: Given IV and PO
  Double-Unit Umbilical Cord Blood Transplantation: Undergo double-unit UCBT
  Fludarabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV and PO
  Total-Body Irradiation: Undergo high-dose or moderate-intensity TBI
  Umbilical Cord Blood Transplantation: Undergo UCBT
  Thiotepa: Given IV
Period: Overall Study
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa
Started | 108 | 27
Started: Single-cord Transplant | 34 | 17
Started: Double-cord Transplant | 74 | 10
Completed: Single-cord Transplant | 26 | 10
Completed: Double-cord Transplant | 48 | 5
Completed | 74 | 15
Not Completed | 34 | 12
Not completed — Death | 24 | 9
Not completed — Relapse | 8 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide: Patients enrolled to receive myeloablative conditioning comprising fludarabine IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 and -6, and undergo high-dose TBI BID on days -4 to -1. Patients then undergo single- or double-unit UCBT on day 0.
  Patients to receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Cyclophosphamide: Given IV
  Cyclosporine: Given IV and PO
  Fludarabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV and PO
  Total-Body Irradiation: Undergo high-dose TBI
  Umbilical Cord Blood Transplantation: Undergo UCBT (either single- or double-cord)
- Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa: Patients enrolled to receive myeloablative conditioning comprising fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 2-4 hours on days -5 and -4, and middle-intensity TBI QD on days -2 and -1. Patients then undergo single- or double-unit UCBT on day 0.
  Patients to receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Cyclophosphamide: Given IV
  Cyclosporine: Given IV and PO
  Fludarabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV and PO
  Total-Body Irradiation: Undergo moderate-intensity TBI
  Umbilical Cord Blood Transplantation: Undergo UCBT (either single- or double-cord)
  Thiotepa: Given IV
- Total: Total of all reporting groups
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa | Total
Number analyzed (Participants) | 108 | 27 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52 | 14 | 66
  Between 18 and 65 years | 56 | 13 | 69
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 22 [0 to 45] | 24.5 [1 to 63] | 22.5 [0 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 14 | 59
  Male | 63 | 13 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 4 | 37
  Not Hispanic or Latino | 73 | 23 | 96
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 4 | 1 | 5
  White | 68 | 17 | 85
  More than one race | 6 | 1 | 7
  Unknown or Not Reported | 16 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival defined as patient being alive at 1 year post-transplant. Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: 1 year post-transplant
Population: Analysis population is all patients who underwent UCB transplant on study, whether completed treatment on study or relapsed at later timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant: Patients receive myeloablative conditioning comprising fludarabine IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 and -6, and undergo high-dose TBI BID on days -4 to -1. Patients then undergo single-unit UCBT on day 0.
  Fludarabine: Given IV Cyclophosphamide: Given IV Total-Body Irradiation: Undergo high-dose TBI Umbilical Cord Blood Transplantation: Undergo UCBT
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Cyclosporine: Given IV and PO Mycophenolate Mofetil: Given IV and PO Laboratory Biomarker Analysis: Correlative studies
- Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant: Patients receive myeloablative conditioning comprising fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 2-4 hours on days -5 and -4, and middle-intensity TBI QD on days -2 and -1. Patients then undergo single-unit UCBT on day 0.
  Fludarabine: Given IV Cyclophosphamide: Given IV Thiotepa: Given IV Total-Body Irradiation: Undergo moderate-intensity TBI Umbilical Cord Blood Transplantation: Undergo UCBT
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Cyclosporine: Given IV and PO Mycophenolate Mofetil: Given IV and PO Laboratory Biomarker Analysis: Correlative studies
- Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant: Patients receive myeloablative conditioning comprising fludarabine IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 and -6, and undergo high-dose TBI BID on days -4 to -1. Patients then undergo double-unit UCBT on day 0.
  Fludarabine: Given IV Cyclophosphamide: Given IV Total-Body Irradiation: Undergo high-dose TBI Umbilical Cord Blood Transplantation: Undergo UCBT
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Cyclosporine: Given IV and PO Mycophenolate Mofetil: Given IV and PO Laboratory Biomarker Analysis: Correlative studies
- Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant: Patients receive myeloablative conditioning comprising fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 2-4 hours on days -5 and -4, and middle-intensity TBI QD on days -2 and -1. Patients then undergo double-unit UCBT on day 0.
  Fludarabine: Given IV Cyclophosphamide: Given IV Thiotepa: Given IV Total-Body Irradiation: Undergo moderate-intensity TBI Umbilical Cord Blood Transplantation: Undergo UCBT
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour every 8 or 12 hours, then cyclosporine PO (if tolerated), on days -3 to 100 with taper on day 101. Patients also receive mycophenolate mofetil IV every 8 hours on days 0 to 7 and then PO (if tolerated) TID on days 8-30. Mycophenolate mofetil is tapered to BID on day 30 or 7 days after engraftment if there is no acute GVHD, and then tapered over 2-3 weeks beginning on day 45 (or 15 days after engraftment if engraftment occurred > day 30) after engraftment if there continues to be no evidence of acute GVHD.
  Cyclosporine: Given IV and PO Mycophenolate Mofetil: Given IV and PO Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 33 | 17 | 72 | 10
Participants | 28 | 15 | 53 | 7

2. Secondary Outcome: Change in Level of Chimerism at Multiple Time Points
Description: Peripheral blood chimerism studies (sorted for CD3, CD14, CD33, CD56 cells) were collected for all UCBT recipients for days 28, 56, 80, 365, and 730 post-transplant. The combined median of the percent donor, along with full range, is captured to show change in level of chimerism at multiple time points up to 2 years post-transplant. Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: Baseline up to 2 years post-transplant
Population: Participants who received UCBT on study with chimerism data available within window as specified in protocol.
Measure: Median (Full Range); unit: percentage chimerism (%)
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 33 | 17 | 72 | 10
percentage chimerism (%)
  Combined median of CD3 at days (24, 56, 80, 180, 365, 730) | 100 [44 to 100] | 100 [69 to 100] | 100 [67 to 100] | 100 [88 to 100]
  Combined median of CD14 at days (24, 56, 80, 180, 365, 730) | 100 [0 to 100] | 100 [100 to 100] | 100 [91 to 100] | 100 [100 to 100]
  Combined median of CD33 at days (24, 56, 80, 180, 365, 730) | 100 [99 to 100] | 100 [98 to 100] | 100 [50 to 100] | 100 [91 to 100]
  Combined median of CD56 at days (24, 56, 80, 180, 365, 730) | 100 [0 to 100] | 100 [100 to 100] | 100 [60 to 100] | 100 [90 to 100]

3. Secondary Outcome: Incidence of Transplant-related Mortality (TRM)
Description: Defined as death due to complication (other than relapse) within 6 months following UCBT. Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: At 6 months post-transplant
Population: Analysis population is all patients who underwent UCB transplant on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 33 | 17 | 72 | 10
Participants | 2 | 1 | 9 | 1

4. Secondary Outcome: Neutrophil Engraftment
Description: Neutrophil engraftment after UCBT is defined as the first day of absolute neutrophil count (ANC) ≥ 5 x 10⁸/L for 3 consecutive measures. Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: Up to day 42 post-transplant
Population: Analysis population is all patients who underwent UCB transplant and experienced ANC engraftment by day 42 post-transplant on study. 4 patients did engraft ANC after day 42 post-transplant, but are not included in this analysis due to protocol definition of engraftment period.
Measure: Median (Full Range); unit: Days post-transplant
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 30 | 16 | 65 | 8
Days post-transplant | 19 [12 to 42] | 19 [13 to 40] | 22 [12 to 39] | 20 [15 to 29]

5. Secondary Outcome: Platelet Engraftment
Description: Platelet (PLT) engraftment after UCBT is defined as the first day of platelet count > 20,000/μl without subsequent transfusions for 7 days. Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: Up to 6 months post-transplant
Population: Analysis population is all patients who underwent UCB transplant and experienced PLT engraftment by 6 months post-transplant on study.
Measure: Median (Full Range); unit: Days post-transplant
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 29 | 16 | 60 | 8
Days post-transplant | 34 [21 to 82] | 35 [18 to 90] | 41 [22 to 158] | 37 [30 to 56]

6. Secondary Outcome: Event of Grade II-IV and III-IV Acute Graft-versus-host Disease (aGVHD)
Description: Each event of aGVHD will be assigned an overall aGVHD score based on extent of skin rash, volume of diarrhea, and maximum bilirubin level, per protocol Appendix I, "GVHD Staging and Grading." Scores reported range from most mild at 2, to worse at 4. Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: Up to day 100 post-transplant
Population: Participants who received UCBT on study.
Measure: Number; unit: events
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 33 | 17 | 72 | 10
events
  Grade II-IV aGVHD | 29 | 14 | 51 | 5
  Grade III-IV aGVHD | 7 | 2 | 17 | 1

7. Secondary Outcome: Event of Chronic Graft-verses-host-disease (cGVHD)
Description: Each event of cGVHD level will be assessed overall as either 'Limited' (mild and with single organ involvement) or 'Extensive' (involvement of two or more organs with symptoms) based on extent of skin rash, volume of diarrhea, and maximum bilirubin level, per protocol Appendix I, "GVHD Staging and Grading." Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: Up to 2 years post-transplant
Population: Participants who received UCBT on study.
Measure: Number; unit: events
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 33 | 17 | 72 | 10
events
  Limited cGVHD | 12 | 6 | 11 | 5
  Extensive cGVHD | 14 | 5 | 44 | 2

8. Secondary Outcome: Event of Clinically Significant Infections
Description: Each event of infection will be assessed to determine whether or not it is clinically significant. An infection is defined as clinically significant when it is scored as ≥ grade 3 (where worse outcomes are associated with higher grading) in accordance with the CTCAE version 3.0/protocol Appendix VI, and constitutes a Serious Adverse Event (SAE). Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: Up to 2 years post-transplant
Population: Participants who received UCBT on study.
Measure: Number; unit: events
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 33 | 17 | 72 | 10
events | 2 | 0 | 21 | 1

9. Secondary Outcome: Incidence of Relapse
Description: Relapse is defined as post-transplant disease recurrence in participants who had initially recovered or improved, with incidence measured from Day 0 to 1 year post-transplant, and from 1 year post-transplant to 2 years post-transplant. Monitoring will take place separately for the single and double UCBT cohorts.
Time Frame: At 1 and 2 years post-transplant
Population: Analysis population is all patients who underwent UCB transplant on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 33 | 17 | 72 | 10
Participants
  Relapse at 1 year | 2 | 4 | 11 | 0
  Relapse at 2 year | 0 | 0 | 0 | 1
  No relapse while on study | 31 | 13 | 61 | 9

10. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time (in days) from UCBT until the disease progresses or the patient dies from any cause, with incidence measured up to 2 years post-transplant. Monitoring will take place separately for the single and double UCBT cohorts. Measure will be reported as the median amount of days from full minimum and maximum range.
Time Frame: Up to 2 years post-transplant
Population: Analysis population is all patients who underwent UCB transplant on study.
Measure: Median (Full Range); unit: Days post-transplant
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Single-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Single-cord Transplant | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide; Double-cord Transplant | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa; Double-cord Transplant
Number analyzed (Participants) | 33 | 17 | 72 | 10
Days post-transplant | 167 [90 to 181] | 155 [32 to 194] | 112 [6 to 353] | 317 [55 to 724]

ADVERSE EVENTS:
Time Frame: Grade 3 or 4 (or highly unusual grade 2) adverse events were monitored, assessed, and collected from the start of study treatment (pre-transplant conditioning) through Day +100 post-transplant. All-Cause Mortality was monitored/assessed from the start of study treatment (pre-transplant conditioning) up to 2 years post-transplant. If a patient experiences relapse or graft failure and goes on to further treatment off protocol, adverse events are no longer collected with the exception of death.
Description: For the purpose of this study, hospitalizations for protocol-scheduled procedures, blood product transfusions, or for social reasons (i.e., awaiting transport home) will not be considered serious adverse events. Hospitalization will be considered a serious adverse event (SAE) if it is unexpected or the duration of the hospital stay is unexpected. Otherwise, the definition of adverse event and/or serious adverse event aligns with the clinicaltrials.gov definitions.
Arm/Group | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa
All-Cause Mortality (participants affected / at risk) | 24/108 | 9/27
Serious Adverse Events (participants affected / at risk) | 47/108 | 7/27
Other Adverse Events (participants affected / at risk) | 73/108 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide (N=108) | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa (N=27)
Acute kidney injury (AKI) (Renal and urinary disorders) | 3 (3) | 1 (1) — A disorder characterized by the acute loss of renal function (within 2 weeks) and is traditionally classified as pre-renal (low blood flow into kidney), renal (kidney damage) and post-renal causes (ureteral or bladder outflow obstruction).
Renal failure (Renal and urinary disorders) | 3 (3) | 2 (2) — Chronic dialysis or renal transplant indicated.
Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) — Acute respiratory distress syndrome (ARDS) is a serious lung condition that causes fluid to build up in the lungs, making it difficult to breathe and get oxygen into the body. Graded on whether intubation is indicated.
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — Grade 4 hyperbilirubinemia is bilirubin level raised by >10.0 times the Upper Limit Number (ULN)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 1 (1) | 0 (0) — Loss of heart activity due to irregular heart rhythm. Life-threatening.
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Inflammation of the gallbladder. Interventional radiology, endoscopic, or operative intervention indicated.
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) — Confusion or delirium interfering with activities of daily living (ADLs).
Diarrhea (Gastrointestinal disorders) | 9 (9) | 0 (0) — Increase of ≥7 stools per day over baseline; incontinence; IV fluids ≥24 hrs; hospitalization; severe increase in output compared to baseline; interfering with ADL.
Encephalopathy (Nervous system disorders) | 3 (3) | 2 (2) — Cognitive disturbance; depressed level of consciousness. Grade 3= signs or symptoms interfering with ADL; hospitalization indicated. Grade 4= life-threatening or disabling.
Syncope (fainting) (Nervous system disorders) | 2 (2) | 0 (0) — A brief loss of consciousness that is followed by a quick and complete recovery.
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 109/L, fever ≥38.5°C).
Pain - Select: Head/headache (Nervous system disorders) | 1 (1) | 0 (0) — Headache causing severe pain; pain or analgesics severely interfering with ADL.
Hemorrhage, pulmonary/ upper respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — Bronchopulmonary hemorrhage. Grade 3=Transfusion, interventional radiology, endoscopic, or operative intervention indicated; radiation therapy. Grade 4=Life-threatening consequences; major urgent intervention indicated.
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — Grade 4= Potassium at a level >7.0 mmol/L.
Hypertension (Vascular disorders) | 3 (4) | 0 (0) — Grade 3=Raised blood pressure with symptoms, requiring more than one drug or more intensive therapy than previously. Grade 4=Life-threatening consequences (e.g., hypertensive crisis).
Hypotension (Vascular disorders) | 4 (7) | 1 (2) — Low blood pressure, symptomatic; Grade 3=Sustained (≥24 hrs) therapy, resolves without persisting physiologic consequences. Grade 4=Shock (e.g., acidemia; impairment of vital organ function).
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (8) — A disorder characterized by a decrease in the level of oxygen in the body. Grade 3=Decreased O2 saturation at rest; continuous oxygen indicated. Grade 4=Life-threatening; intubation or ventilation indicated. Grade 5=respiratory failure/death.
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 8 (9) | 1 (1) — A disorder characterized by an infectious process involving the lungs, including pneumonia. IV antibiotic, antifungal, or antiviral intervention indicated; invasive intervention indicated.
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 6 (7) | 0 (0) — Also called sepsis; disorder characterized by the presence of pathogenic microorganisms in the blood stream that cause a rapidly progressing systemic reaction that may lead to shock. Blood culture positive with signs or symptoms; treatment indicated.
Infection with Grade 3 or 4 neutrophils - Bladder or urinary tract (Infections and infestations) | 4 (4) | 0 (0) — Infection documented clinically or microbiologically with ANC <1.0 x 10^9/L. A disorder characterized by an infectious process involving the bladder or urinary tract.
Infection with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 1 (1) | 0 (0) — Infection documented clinically or microbiologically with ANC <1.0 x 10^9/L. Sepsis; disorder characterized by the presence of pathogenic microorganisms in the blood stream that cause a rapidly progressing systemic reaction that may lead to shock.
Acute infusion reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — A disorder characterized by adverse reaction to the infusion of pharmacological or biological substances.
Hemorrhage, GI - Abdominal NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) — Transfusion, interventional radiology, endoscopic, or operative intervention indicated; radiation therapy. Life-threatening consequences; major urgent intervention indicated.
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — A disorder characterized by abnormally high acidity (high hydrogen-ion concentration) of the blood and other body tissues. Grade 4=pH <7.3 with life-threatening consequences.
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) — A disorder characterized by new or increased apprehension of danger and dread accompanied by restlessness, tension, tachycardia, and dyspnea unattached to a clearly identifiable stimulus.
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 4 (4) | 1 (1) — A serious medical emergency that occurs when two or more organ systems in the body are no longer working properly. Grade 5 is the only appropriate grade.
Myelitis (Infections and infestations) | 0 (0) | 1 (1) — A disorder characterized by inflammation involving the spinal cord. Symptoms include weakness, paresthesia, sensory loss, marked discomfort and incontinence.
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — A disorder characterized by necrotic changes in the bone tissue due to interruption of blood supply. Most often affecting the epiphysis of the long bones, the necrotic changes result in the collapse and the destruction of the bone structure.
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1) | 0 (0) — A disorder characterized by fluid collection within the pericardial sac, usually due to inflammation.
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1 (1) | 0 (0) — Death resulting from a recurrence of disease in sites other than the bone marrow. Grade 5 is the only appropriate grade.
Infection with normal ANC - Throat/lymph nodes (retropharyngeal abscess) (Infections and infestations) | 1 (1) | 0 (0) — A retropharyngeal abscess is a pus-filled collection in the back of the throat that can be life-threatening. It's caused by a bacterial infection in the lymph nodes behind the throat, which are part of the immune system.
Seizure (Nervous system disorders) | 3 (3) | 2 (3) — A disorder characterized by a sudden, involuntary skeletal muscular contractions of cerebral or brain stem origin.
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 3 (3) | 0 (0) — A disorder characterized by severe hepatic injury as a result of the blood vessels of the liver becoming inflamed and/or blocked.
Supraventricular and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) — A disorder characterized by a dysrhythmia with a heart rate less than 60 beats per minute that originates in the sinus node. Symptomatic; intervention indicated.
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0) — A disorder characterized by inadequate absorption of nutrients in the small intestine. Symptoms include weight loss, abdominal marked discomfort, bloating and diarrhea.
Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura [TTP] (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — A disorder characterized by the presence of microangiopathic hemolytic anemia, thrombocytopenic purpura, fever, renal abnormalities and neurological abnormalities such as seizures, hemiplegia, and visual disturbances. An acute or subacute condition.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: High-dose TBI + Fludarabine + Cyclophosphamide (N=108) | Regimen B: Middle-intensity TBI + Fludarabine + Cyclophosphamide + Thiotepa (N=27)
Allergic reaction/hypersensitivity (Immune system disorders) | 2 (2) | 1 (1) — Urticaria with manifestations of allergic or hypersensitivity reaction is graded as Allergic reaction/hypersensitivity (including drug fever).
Febrile neutropenia (Blood and lymphatic system disorders) | 33 (50) | 14 (14) — Fever of unknown origin without clinically or microbiologically documented infection; ANC <1.0 x 109/L, fever ≥38.5°C.
CD4 count (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — CD4 count <50/mm3 <0.05 x 109 /L.
Leukocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Leukocyte (total WBC) count <1000/mm3 <1.0 x 109 /L.
Hemolysis (Blood and lymphatic system disorders) | 5 (5) | 0 (0) — e.g., immune hemolytic anemia, drug-related hemolysis
Iron overload (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2) | 2 (3)
Prolonged QTc interval (Cardiac disorders) | 1 (1) | 2 (3)
Cardiac General - Other (Heart failure) (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 13 (15) | 11 (13)
Hypotension (Blood and lymphatic system disorders) | 10 (12) | 4 (5)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Coagulation, Other (Coagulopathy) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombotic microangiopathy (TMA) (Blood and lymphatic system disorders) | 3 (3) | 1 (1) — e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS]
Fatigue (General disorders) | 2 (2) | 1 (1)
Insomnia (General disorders) | 1 (2) | 0 (0)
Fever (General disorders) | 3 (3) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 59 (77) | 11 (13)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Mucositis (Gastrointestinal disorders) | 32 (55) | 9 (9)
Acute kidney injury (AKI) (Renal and urinary disorders) | 2 (2) | 3 (4)
Alanine aminotransferase (ALT) increased, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 (6) | 0 (0)
Anorexia (Gastrointestinal disorders) | 9 (10) | 5 (6)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (AST) (Investigations) | 2 (3) | 0 (0)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperbilirubinemia (Investigations) | 10 (14) | 3 (3)
Cytomegalovirus virus (CMV) reactivation (Infections and infestations) | 5 (9) | 4 (4)
Cystitis (Renal and urinary disorders) | 1 (3) | 0 (0)
Thrombosis/thrombus/ embolism (Vascular disorders) | 1 (1) | 0 (0) — e.g. Deep vein thrombosis
Mood alteration - Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (18) | 5 (5)
Disseminated Adenovirus (ADV) (Infections and infestations) | 6 (9) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Renal/Genitourinary, Other (Veno-occlusive disease [VOD]) (Renal and urinary disorders) | 3 (4) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hemorrhage/bleeding (General disorders) | 8 (9) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (17) | 4 (5)
Infection in blood (Infections and infestations) | 44 (70) | 7 (10)
Infection in urinary tract (urinary tract infection; UTI) (Infections and infestations) | 12 (16) | 0 (0)
Infection in respiratory tract (Infections and infestations) | 13 (18) | 4 (4) — e.g. pneumonia, RSV, etc.
Infection in gastrointestinal tract (Infections and infestations) | 6 (8) | 3 (3) — e.g. colitis infectious, enterocolitis infectious, C. Diff, etc.
Infection, Other (Infections and infestations) | 10 (10) | 1 (1) — e.g. skin/cellulitis, cerebral spinal fluid (CSF), mucosal (mouth, perianal, etc.), sinus/sinusitis, etc.
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Distention/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Irritable bowel syndrome (IBS) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-organ failure (MOF) (General disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neutrophil count (ANC) decreased (Investigations) | 1 (1) | 2 (4) — Captured when occurring after post-transplant engraftment after post-transplant engraftment
Pain, Other - Bone pain (General disorders) | 1 (3) | 0 (0)
Pain (General disorders) | 5 (14) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Weight gain (General disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study initiated in 2005, but Arm B was added to the study design in 2019. Therefore patient accrual in Arm B is lower than Arm A, though rate of accrual was comparable once both arms were available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT00719888/Prot_SAP_000.pdf
  • Informed Consent Form: Regimen A ICF (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT00719888/ICF_001.pdf
  • Informed Consent Form: Regimen B ICF (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT00719888/ICF_002.pdf